CLINICAL TRIAL: NCT01524614
Title: Effect of Continuous Positive Airway Pressure Ventilation Through Nasal Mask on Upper Airway Patency During Induction of Anesthesia
Brief Title: Safety Study of Continuous Positive Airway Pressure Via a Nasal Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yandong Jiang, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2010p002823
Record Dates: First submitted 2012-01-12; First posted 2012-02-02 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Upper Airway Obstruction
Keywords: continuous positive airway pressure; nasal mask; upper airway obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nasal mask with no PEEP (Experimental): Nasal mask with PEEP 0, then add PEEP 5, and 10
  Interventions: Procedure: nasal mask
- Nasal mask with PEEP (Experimental): Nasal mask with PEEP 5, then add PEEP 10
  Interventions: Procedure: nasal mask
- Face mask with no PEEP (Experimental): Face mask with PEEP 0 then add PEEP 5, 10
  Interventions: Procedure: nasal mask
- Face mask with PEEP (Experimental): Face mask with PEEP 5, then add PEEP 10
  Interventions: Procedure: nasal mask

INTERVENTIONS:
Procedure: nasal mask — nasal mask use instead of face mask

SUMMARY:
Upper airway obstruction (UAO) is common complication during induction of general anesthesia. The mechanism of UAO during anesthesia has not been well understood. Posterior displacement of soft palate are believed to be the primary contributing factors. The mechanism of UAO during anesthesia share many similarities with obstructive sleep apnea (OSA). Since nasal continuous positive airway pressure (nCPAP) can maintain the airway patent in patients with OSA, the investigators hypothesize that nCPAP during induction of anesthesia will reduce the incidence and severity of UAO.

ELIGIBILITY:
Inclusion Criteria:

Patients,between 18-65 years of age meeting ASA physical status classification I-II requiring general anesthesia for elective surgery who are able to breathe through both their nose and mouth while awake.

Exclusion Criteria:

1. Patients with major cardiovascular disease, respiratory disease, cerebral vascular disease or American Society of Anesthesiologists physical status class III or greater.
2. Abnormal vital signs on the day of admission for surgery [heart rate (HR, > 100 bpm or < 40 bpm), blood pressure (BP, > 180/100 mmHg or < 90/60 mmHg), room air transcutaneous oxyhemoglobin saturation (SPO2) < 96%] that are not correctable with his or her routine medication or commonly used pre-operative medication.
3. Unable to open mouth (< 2.5 cm) or unable to breathe through their mouth or nose.
4. Subjects with a beard, an abnormal facial structure or other factors precluding obtaining a viable face mask fit without air leak. Also, subjects having claustrophobia that can not tolerate the mask.
5. Any person with an anticipated difficult airway. This will include subjects who require or may require either a fiberoptic intubation or intubation while awake and subjects with known OSA or body mass index (BMI) greater than 35 km/m2.
6. Gastric-esophageal reflex or a full stomach.
7. The subject has remained in bed for more than 24 hours.
8. Neurological symptoms associated with neck extension, a neurological deficit from a previous stroke or spinal cord injury, a recent stroke or transient ischemic attack (TIA) within 2 weeks.
9. Pregnant women and women less than one month post-partum. Ruling out pregnancy will be conducted by careful history and physical examination as performed routinely prior to surgery. If the history is believed to be unreliable, the patient will be excluded unless a pregnancy test is performed and the result of the test is negative.
10. Emergency cases and subjects who have not adhered to the ASA NPO (Nil Per Os) guidelines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
expired tidal volume | Average of one minute after anesthesia induction
  Estimated time from induction of anesthesia (drugs given for anesthesia induction) to apnea is one minute.

SECONDARY OUTCOMES:
volume of CO2 | Average of one minute after anesthesia induction
  Estimated time from induction of anesthesia (drugs given for anesthesia induction) to apnea is one minute.

CONTACTS AND LOCATIONS:
Overall Officials: Yandong Jiang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Anesthesia and Critical Care, Mass General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Oto J, Li Q, Kimball WR, Wang J, Sabouri AS, Harrell PG, Kacmarek RM, Jiang Y. Continuous positive airway pressure and ventilation are more effective with a nasal mask than a full face mask in unconscious subjects: a randomized controlled trial. Crit Care. 2013 Dec 23;17(6):R300. doi: 10.1186/cc13169. PMID 24365207